CLINICAL TRIAL: NCT05105139
Title: Retrospective Study to Evaluate the Safety of Sebryl® and / or Sebryl Plus® in the Treatment of Seborrheic Dermatitis and Psoriasis of the Scalp in Routine Medical Practice.
Brief Title: Study to Evaluate the Safety of Sebryl® and Sebryl Plus® in Seborrheic Dermatitis and Psoriasis of Scalp
Status: Completed | Type: Observational
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: SIL-31103-IV-21(1)
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Seborrheic Dermatitis; Psoriasis of Scalp
Keywords: Allantoin; Coal Tar; Clioquinol; Triclosan; Seborrheic Dermatitis; Psoriasis of Scalp
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Allantoin; Coal Tar; Clioquinol; Triclosan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A1: Allantoin / Coal Tar / Clioquinol (Sebryl®): Pharmaceutical Form: Shampoo Dosage: 0.2 g/ 5.0 g/ 3.0 g Administration way: For scalp use
  Interventions: Other: Allantoin/ Coal Tar/ Clioquinol
- A2: Allantoin/ Coal Tar/ Clioquinol/ Triclosan (Sebryl Plus®): Pharmaceutical Form: Shampoo Dosage: 0.2 g/ 3.0 g/ 3.0 g/ 0.3 g Administration way: For scalp use
  Interventions: Other: Allantoin/ Coal Tar/ Clioquinol/ Triclosan

INTERVENTIONS:
Other: Allantoin/ Coal Tar/ Clioquinol — Pharmaceutical Form: Shampoo Dosage: Allantoin 0.2 g/ Coal Tar 5.0 g/ Clioquinol 3.0 g Administration way: For scalp use
  Other Names: Sebryl®
  Groups: A1: Allantoin / Coal Tar / Clioquinol (Sebryl®)
Other: Allantoin/ Coal Tar/ Clioquinol/ Triclosan — Pharmaceutical Form: Shampoo Dosage: Allantoin 0.2 g/ Coal Tar 3.0 g/ Clioquinol 3.0 g/ Triclosan 0.3 g. Administration way: For scalp us
  Other Names: Sebryl Plus®
  Groups: A2: Allantoin/ Coal Tar/ Clioquinol/ Triclosan (Sebryl Plus®)

SUMMARY:
Observational, descriptive, retrospective, multicenter study to evaluate the safety of the treatment with Sebryl® and / or Sebryl Plus® in the management of seborrheic dermatitis and psoriasis of the scalp in routine medical practice.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the frequency and intensity of adverse events presented during treatment with Sebryl® and / or Sebryl Plus® for the management of seborrheic dermatitis and psoriasis of the scalp. The sample will be at convenience. The files of the patients who have received treatment with Sebryl® and / or Sebryl Plus® in the last 5 years (2016 to 2021) will be chosen.

The researchers or the personnel designated by them will capture the information recorded by the treating physicians in the clinical file, sociodemographic, clinical and safety data that were presented after the prescription of Sebryl® and / or Sebryl Plus®.

ELIGIBILITY:
Inclusion Criteria:

* Any sex.
* Treatment with Sebryl® and / or Sebryl Plus® documented, for at least 2 consultations.
* That the patient has been questioned about possible adverse events

Exclusion Criteria:

* That the patient has used some other concomitant treatment for seborrheic dermatitis and psoriasis on the scalp.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of indistinct sex with seborrheic dermatitis and / or psoriasis of the scalp who, according to medical criteria, have been candidates for treatment with Sebryl® and / or Sebryl Plus®.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Proportion of adverse events | Last 5 years
  Evaluate the presence or absence of adverse events reported in the clinical files.
Classify adverse events | Last 5 years
  Classify reported adverse events according to seriousness, severity (intensity) and causality of the clinical manifestation
Mean age in years | Last 5 years
  Describe the mean age in years of the patients included in the study.
Describe study population by gender ratio | Last 5 years
  Describe the proportion of women and men included in the study
Describe the body mass index through weight and heigh | Last 5 years
  Describe the body mass index of the study population calculated through weight and heigh of the patient and using the formula kilogram over square meter.
Describe the blood pressure millimetres of mercury (mmHg) | Last 5 years
  Describe the blood pressure in mmHg of the patients included in the study.
Mean heart rate in beats per minute | Last 5 years
  Describe the mean heart rate in beats per minute of the patients included in the study.
Percentage of times use outside of expected indications | Last 5 years
  Percentage of times Sebryl® and / or Sebryl® Plus were used outside of expected indications.

SECONDARY OUTCOMES:
Description of usage pattern according to prescribed dosage | Last 5 years
  Describe according to prescribed dosage the pattern of use of Sebryl® and / or Sebryl Plus® in the management of seborrheic dermatitis and psoriasis of the scalp.
Description of usage pattern according to prescribed time | Last 5 years
  Describe according to prescribed time the pattern of use of Sebryl® and / or Sebryl Plus® in the management of seborrheic dermatitis and psoriasis of the scalp.

CONTACTS AND LOCATIONS:
Overall Officials: María E Morales Barrera, M.D, Principal Investigator — Independent consultant
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christophers E. Psoriasis--epidemiology and clinical spectrum. Clin Exp Dermatol. 2001 Jun;26(4):314-20. doi: 10.1046/j.1365-2230.2001.00832.x. PMID 11422182
- [Background] Parisi R, Symmons DP, Griffiths CE, Ashcroft DM; Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol. 2013 Feb;133(2):377-85. doi: 10.1038/jid.2012.339. Epub 2012 Sep 27. PMID 23014338
- [Background] Gibbs S. Skin disease and socioeconomic conditions in rural Africa: Tanzania. Int J Dermatol. 1996 Sep;35(9):633-9. doi: 10.1111/j.1365-4362.1996.tb03687.x. PMID 8876289
- [Background] Rachakonda TD, Schupp CW, Armstrong AW. Psoriasis prevalence among adults in the United States. J Am Acad Dermatol. 2014 Mar;70(3):512-6. doi: 10.1016/j.jaad.2013.11.013. Epub 2014 Jan 2. PMID 24388724
- [Background] Danielsen K, Olsen AO, Wilsgaard T, Furberg AS. Is the prevalence of psoriasis increasing? A 30-year follow-up of a population-based cohort. Br J Dermatol. 2013 Jun;168(6):1303-10. doi: 10.1111/bjd.12230. PMID 23374051
- [Background] Rendon A, Schakel K. Psoriasis Pathogenesis and Treatment. Int J Mol Sci. 2019 Mar 23;20(6):1475. doi: 10.3390/ijms20061475. PMID 30909615
- [Background] Ortonne J, Chimenti S, Luger T, Puig L, Reid F, Trueb RM. Scalp psoriasis: European consensus on grading and treatment algorithm. J Eur Acad Dermatol Venereol. 2009 Dec;23(12):1435-44. doi: 10.1111/j.1468-3083.2009.03372.x. Epub 2009 Jul 15. PMID 19614856
- [Background] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Background] Sommer DM, Jenisch S, Suchan M, Christophers E, Weichenthal M. Increased prevalence of the metabolic syndrome in patients with moderate to severe psoriasis. Arch Dermatol Res. 2006 Dec;298(7):321-8. doi: 10.1007/s00403-006-0703-z. Epub 2006 Sep 22. PMID 17021763
- [Background] Gerdes S, Mrowietz U, Boehncke WH. [Comorbidity in psoriasis]. Hautarzt. 2016 Jun;67(6):438-44. doi: 10.1007/s00105-016-3805-3. German. PMID 27221798
- [Background] Krueger G, Koo J, Lebwohl M, Menter A, Stern RS, Rolstad T. The impact of psoriasis on quality of life: results of a 1998 National Psoriasis Foundation patient-membership survey. Arch Dermatol. 2001 Mar;137(3):280-4. PMID 11255325
- [Background] Nast A, Kopp IB, Augustin M, Banditt KB, Boehncke WH, Follmann M, Friedrich M, Huber M, Kahl C, Klaus J, Koza J, Kreiselmaier I, Mohr J, Mrowietz U, Ockenfels HM, Orzechowski HD, Prinz J, Reich K, Rosenbach T, Rosumeck S, Schlaeger M, Schmid-Ott G, Sebastian M, Streit V, Weberschock T, Rzany B; Deutsche Dermatologische Gesellschaft (DDG); Berufsverband Deutscher Dermatologen (BVDD). Evidence-based (S3) guidelines for the treatment of psoriasis vulgaris. J Dtsch Dermatol Ges. 2007 Jul;5 Suppl 3:1-119. doi: 10.1111/j.1610-0387.2007.06172.x. PMID 17615051
- [Background] Pardasani AG, Feldman SR, Clark AR. Treatment of psoriasis: an algorithm-based approach for primary care physicians. Am Fam Physician. 2000 Feb 1;61(3):725-33, 736. PMID 10695585
- [Background] Borda LJ, Wikramanayake TC. Seborrheic Dermatitis and Dandruff: A Comprehensive Review. J Clin Investig Dermatol. 2015 Dec;3(2):10.13188/2373-1044.1000019. doi: 10.13188/2373-1044.1000019. Epub 2015 Dec 15. PMID 27148560
- [Background] Langner A, Wolska H, Hebborn P. Treatment of psoriasis of the scalp with coal tar gel and shampoo preparations. Cutis. 1983 Sep;32(3):290-1, 295-6. PMID 6627992
- [Background] Puig L, Ribera M, Hernanz JM, Belinchon I, Santos-Juanes J, Linares M, Querol I, Colome E, Caballe G. [Treatment of scalp psoriasis: review of the evidence and Delphi consensus of the Psoriasis Group of the Spanish Academy of Dermatology and Venereology]. Actas Dermosifiliogr. 2010 Dec;101(10):827-46. Spanish. PMID 21159259